CLINICAL TRIAL: NCT05802329
Title: A Phase 1 Study To Assess The Safety And Efficacy Of OCU200 For Center-Involved Diabetic Macular Edema
Brief Title: Phase I Study to Assess the Safety and Efficacy of OCU200 for Center-Involved Diabetic Macular Edema (DME)
Acronym: DME
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OCU200-101
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Center Involved Diabetic Macular Edema; Diabetic Macular Edema
Keywords: anti-VEGF; Transferrin; Tumstatin; DME

STUDY DESIGN:
Intervention Model Description: 3+3 design with parallel and sequential dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 3+3 participants will receive intravitreal injection of OCU200 (0.5 mg/mL concentration).
  Interventions: Drug: OCU200
- Cohort 2 (Experimental): 3+3 participants will receive intravitreal injection of OCU200 (1 mg/ML concentration).
  Interventions: Drug: OCU200
- Cohort 3 (Experimental): 3+3 participants will receive intravitreal injection of OCU200 (2 mg/mL concentration).
  Interventions: Drug: OCU200
- Cohort 4 (Experimental): 3+3 participants will receive intravitreal injection of OCU200 (5 mg/mL concentration).
  Interventions: Drug: OCU200

INTERVENTIONS:
Drug: OCU200 — Intravitreal Injection

SUMMARY:
A Phase 1 study to assess the safety and efficacy of OCU200 for center-involved diabetic macular edema

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose ranging study with 4 cohorts in the dose-escalation portion of the study. An accelerated 3+3 design with parallel and sequential dosing will be used.

Under the escalation design, 12 subjects will be enrolled if there are no DLTs and up to 24 subjects under the condition that exactly 1 of the 3 subjects of every cohort if determined to have a DLT.

Each subject will receive a total of 2 intravitreal injections of OCU200 6 weeks apart.

The DSMB will review the sentinel subject 1 week safety data post dosing in every cohort of all 3 subjects.

Cohort 1: 3+3 participants will receive intravitreal injection of OCU200.

Cohort 2: 3+3 participants will receive intravitreal injection of OCU200.

Cohort 3: 3+3 participants will receive intravitreal injection of OCU200.

Cohort 4: 3+3 participants will receive intravitreal injection of OCU200.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 1 or Type 2 Diabetes Mellitus
2. Decreased visual acuity attributable primarily to DME
3. Central-involved DME with central retinal subfield thickness (CST) values, as assessed with spectral-domain optical coherence tomography (SD-OCT) of:

   1. ≥ 320 but ≤ 450µm if male or ≥ 305 but ≤ 435µm if female on Heidelberg Spectralis
   2. ≥ 305 but ≤ 435µm if male or ≥ 290 but ≤ 420µm if female on Zeiss Cirrus
4. BCVA ≤ 78 and ≥ 24 letters on ETDRS chart
5. Sufficient ocular media clarity, pupillary dilation and participant cooperation to permit acquisition of good quality retinal imaging
6. No history of prior anti-VEGF injection or history of at least 2 consecutive intravitreal anti-VEGF injection (less than 7 weeks apart) with incomplete resolution of CST within 1 year.

Note: The last anti-VEGF injection must be administered at least six weeks (45 days) prior to the study treatment (Day 1) in the study eye.

Exclusion Criteria:

1. Presence of any condition that prevent clear visualization of retina (e.g., significant cataract, vitreous hemorrhage)
2. Uncontrolled hypertension
3. Uncontrolled glaucoma
4. Concurrent disease in the study eye, other than central-involved DME
5. Intravitreal or periocular steroid treatment within 3 months prior to the screening visit
6. Any ocular surgery within 3 months prior to the screening visit in the study eye
7. Uncontrolled/poorly controlled diabetes (Glycated hemoglobin (HbA1c) ≥ 10%)
8. History of retinal detachment in the study eye or other retinal vascular disease in the study eye
9. Focal or pan-retinal laser photocoagulation in the study eye within 3 months prior to the screening visit
10. Presence of any inherited retinal disease or history of proliferative diabetic retinopathy
11. History of Renal disease including stage 3b or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Study Drug-related adverse events (SDAE) | 24 weeks
  Counts, frequencies and percentages of SDAEs.
Treatment-emergent adverse events (TEAEs) | 24 weeks
  Counts, frequencies and percentages TEAEs.
Serious adverse events (SAEs) | 24 weeks
  Counts, frequencies and percentages of SAEs.

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) | 24 Weeks (Changes from baseline)
  Measured as the ETDRS letter score on the EVA tester or E-ETDRS charts.
Intraocular pressure (IOP) | 24 weeks(Changes from baseline)
  IOP measurement by applanation or rebound tonometry.
Color fundus photography | 24 Weeks(Changes from baseline)
  Color fundus photographs will be taken to evaluate retinal anatomy and grade diabetic retinopathy severity scale (DRSS).
Spectral Domain Optical Coherence Tomography (SD-OCT) | 24 Weeks(Changes from baseline)
  SD-OCT will be utilized to assess retinal thickness. OCT images and scans will be transmitted to a central reading center for independent analysis.
Spectral Domain Optical Coherence Tomography Angiography (SD-OCTA) | 24 weeks (Changes from baseline)
  SD-OCTA will be utilized to assess retinal vasculature and images will be transmitted to a central reader for independent analysis.
Wide-field Fluorescein Angiography (wf-FA) | 24 weeks (Changes from baseline)
  wf-FA will be conducted at screening and EOS visits to assess central and peripheral vasculature.

OTHER OUTCOMES:
Improvement of diabetic retinopathy severity scale (DRSS) | 24 weeks
  Proportion of participants with ≥ 2-step improvement of diabetic retinopathy severity scale (DRSS)
Change from baseline in BCVA letters. | 24 weeks
  Dose response as assessed by mean change from baseline in BCVA letters and mean number of injections by study visit
Reduction of CST | 24 Weeks
  The proportion of participants having a ≥ 10% reduction of CST at Week 13 and Week 19

CONTACTS AND LOCATIONS:
Overall Officials: Huma Qamar, MD, MPH, CMI, Study Director — Ocugen
Locations (5):
- United States (5):
  - Advanced Research LLC, Deerfield Beach, Florida
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Retina Consultants of Texas Research Centers, Bellaire, Texas
  - Retina Consultants of America, Southlake, Texas
  - Gundersen Health System, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No